CLINICAL TRIAL: NCT04939324
Title: Analyse du Profil moléculaire Des Exosomes de la Veine Pulmonaire Dans le Cancer Bronchique de Stade précoce
Brief Title: Molecular Profiling of Exosomes in Tumor-draining Vein of Early-staged Lung Cancer
Acronym: ExOnSite-Pro
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 87RI20-0067 (ExOnSite-Pro)
Record Dates: First submitted 2021-05-31; First posted 2021-06-25 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Lung Cancer; Exosomes; Non Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood samples at 2 sites: peripheral vein and tumor-draining vein (Other): D0: surgery (inclusion): oncological lung resection
  * Blood samples at 2 sites: peripheral vein and tumor-draining vein
  * Resected tumor analysis Standard clinical and radiological follow-up during 2 years (medical consultation or phone call)
  Interventions: Biological: Blood samples at 2 sites: peripheral vein and tumor-draining vein

INTERVENTIONS:
Biological: Blood samples at 2 sites: peripheral vein and tumor-draining vein — D0: surgery (inclusion): oncological lung resection
  * Blood samples at 2 sites: peripheral vein and tumor-draining vein
  * Resected tumor analysis Standard clinical and radiological follow-up during 2 years (medical consultation or phone call)

SUMMARY:
This is an observational prospective single-center study of 30 patients operated for early-staged non-small cell lung cancer. The main aim is the analysis of molecular profiling of exosome with a sample in tumor-draining vein in order to identify prognostic molecular characteristics associated with cancer recurrence after surgery.

DETAILED DESCRIPTION:
Surgical resection remains the best chance for cure in patients with early-stage non-small-cell lung cancer (NSCLC). Unfortunately, approximately 30-50% of patients will relapse within 5-year of curative surgery despite early TNM-stage. The Identification of prognostic biomarkers of relapse is a necessity. Among them, extracellular vesicles (exosomes) study seems promising in early stage cancers and samples directly in tumor-draining vein to. The pulmonary vein is draining blood directly from the lungs and sampling at this location could provide a higher yield for oncosome. The litterature reports that Navarro et al. are the only team to have link exosome characteristics to oncological outcomes following surgery. The investigators propose to analyze the molecular profiling mediated by these extracellular vesicles in the tumor-draining vein of operated patients.

A peripheral blood sample is recolted before surgery (D-1 or D0). During oncological lung surgery, the pulmonary tumor-drainage vein is first exposed and punctured with a needle prior to subsequent surgical manipulation for resection (D0). A piece of resected tumor will be analyzed for the study (D0). Quantification and size distribution of exosome and molecular cargo of exosome in blood samples (peripheral and pulmonary vein) and tumor are analyzed (DNA sequencing).

Standard clinical and radiological follow-up is then performed and 2-year overall survival and 2-year disease free-survival are checked.

ELIGIBILITY:
Inclusion Criteria:

- Surgical non-small cell lung cancer with pure solid nodule or part-solid ground glass nodule on CT-scan

Exclusion Criteria:

* Pure ground glass nodule,
* Neoadjuvant therapy,
* Second cancer or cancer in the 5 years,
* Pregnancy,
* Patients <18 years-old,
* Tutorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-08-21 (Estimated); Study Completion 2024-06-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate size distribution, concentration and molecular profiling of pulmonary vein exosomes at inclusion | 36 months
  Concentration of extracellular vesicule (million of particule/mL of blood)

SECONDARY OUTCOMES:
Size distribution, molecular profiling of peripheral vein exosome sat inclusion | 36 months
  The size distribution of extracellular vesicules harvested
Mutations and polymorphism in resected lung cancer | 36 months
  Analyze of the molecular profile in the resected tumor tissus
Overall survival | 36 months
  overall survival
Two-year disease-free survival | 24 months
  Two-year disease-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Jérémy Tricard, MD, Principal Investigator — University Hospital, Limoges
Locations (1):
- CHU de Limoges, Limoges, France

IPD SHARING:
Plan to Share IPD: No